CLINICAL TRIAL: NCT02094547
Title: Evaluación Del Efecto de Una Nueva fórmula Infantil Con Ingredientes específicos Sobre el Desarrollo Neurocognitivo e inmunológico en Lactantes
Brief Title: A Neurocognitive and Immunological Study of a New Formula for Healthy Infants
Acronym: COGNIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Laboratorios Ordesa (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: FC0G - 010
Record Dates: First submitted 2014-03-20; First posted 2014-03-24 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Infant Development
Keywords: Infant Formula; Cognition; Neurodevelopment; Immunity; Microbiota
MeSH Terms: interventions — Lactation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- New infant formula (Experimental): New infant formula with key ingredients.
  Interventions: Dietary Supplement: New infant formula
- Standard infant formula (Active Comparator): Standard infant formula
  Interventions: Dietary Supplement: Standard infant formula
- Breastfeeding (Other): Control
  Interventions: Dietary Supplement: Breastfeeding

INTERVENTIONS:
Dietary Supplement: New infant formula — New infant formula
  Arms: New infant formula
Dietary Supplement: Standard infant formula — Standard infant formula
  Arms: Standard infant formula
Dietary Supplement: Breastfeeding — Exclusive breastfeeding or less tan 25% formula intake
  Arms: Breastfeeding

SUMMARY:
To compare the neurocognitive and immunological development in infants fed a new infant formula with functional specific nutrients to infants consuming a standard infant formula.

ELIGIBILITY:
Inclusion Criteria:

* Full-term newborns (>37 weeks and <41 weeks gestation)
* Adequate birth weight for his gestational age (between 3-97 percentiles)
* Inclusion age: from 0 to 2 months (60 days) in the formula fed groups
* Inclusion age: 2-6 months (180 days) in the breastfeeding group
* Maximum 30 days of exclusive breastfeeding in the formula fed groups
* From 30 days on, exclusive or >70% infant formula in the formula fed groups
* Normal Apgar score: 7-10
* Umbilical pH ≥ of 7.10
* Availability to continue during the whole study period
* Informed consent signed ( parent/legal representative)

Exclusion Criteria:

* Participating in other studies.
* Nervous system disorders (hydrocephalic, perinatal hypoxia, intraventricular hemorrhage, neonatal meningitis, septic shock, West Sd...).
* Gastrointestinal disorders (cow's milk protein allergy, lactose intolerance)
* Mother's disease history or during pregnancy: neurological and metabolic diseases, diabetes mellitus type 1, hypothyroidism, undernutrition, infections TORCH complex.
* Mothers receiving anxiolytic or antidepressant treatment during pregnancy or other potentially harmful drug treatments for infants' neurodevelopment.
* Infant's family who in the investigators assessment cannot be expected to comply with the protocol.

Ages: 1 Day to 60 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive Development | At 2nd, 3rd, 4th, 6th, 12th,18th, 30 th months.
  Differences in neurocognitive development inter and intragroup evaluated by visual evoked potential test, general movements test, BAYLEY'S III test, MacArthur test, behavior assessment and cognitive evoked potential test (EEG/ERP).
Neurocognitive Development at 4 and 6 years | At 4 and 6 years of age
  Differences in neurocognitive development evaluated by Computarized battery for neuropsychological evaluation of children, Kaufman Brief Intellligence Test, Language test of Navarre,functional exploration, behavior assessment, questionnaires and cognitive evoked potential test (EEG/ERP).
Neurocognitive Development at 6 years | At 6 years of age
  Functional Magnetic Resonance Image

SECONDARY OUTCOMES:
Formula Tolerability | At 2nd, 3rd, 4th, 6th, 12th and 18th months.
  Evaluation of gastrointestinal symptoms and sleep disorders amongst groups.
Growth | At 2nd, 3rd, 4th, 6th, 12th,18th month; age 2.5, 4 and 6.
  Differences in growth parameters (weight, length, BMI, skin folds, perimeters and z-scores) between groups.
Incidence of infections | At 2nd, 3rd, 4th, 6th, 12th,18th month; age 2.5, 4 and 6.
  Number of infections reported.
Immunoglobulin A secretor (IgAs) levels | At 3rd, 6th, 12th,18th month, and 4 years old.
  Inter and intragroup differences measured by saliva samples analysis.
Impact on microbiota | At 3rd, 6th, 12th and 18th months; 4 and 6 years of age.
  Changes in microbiota composition measured by real-time polymerase chain reaction (RT-PCR) in faeces.
Long Chain Polyunsaturated Fatty Acids (LC-PUFAS) levels | At 3rd, 6th, 12th,18th months; 2.5, 4 and 6 years of age.
  Differences in LC-PUFAS levels inter and intragroup evaluated by oral mucosa samples analysis.
Cardiovascular factors | At 4 and 6 years old
  Blood pressure measurement
Glucose monitoring | At 6 years old
  Urine metabolomic analysis

OTHER OUTCOMES:
Dietary assessment | At 6th, 12th and 18th months; 2.5, 4 and 6 years.
  Food frequency questionnaires and 24 h food recalls.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Campoy, Professor, Principal Investigator — Universidad de Granada
Locations (1):
- Facultad de Medicina, Granada, Spain

REFERENCES:
- [Derived] Dieguez E, Nieto-Ruiz A, Martin-Perez C, Sepulveda-Valbuena N, Herrmann F, Jimenez J, De-Castellar R, Catena A, Garcia-Santos JA, Bermudez MG, Campoy C. Association study between hypothalamic functional connectivity, early nutrition, and glucose levels in healthy children aged 6 years: The COGNIS study follow-up. Front Nutr. 2022 Oct 12;9:935740. doi: 10.3389/fnut.2022.935740. eCollection 2022. PMID 36313089
- [Derived] Cerdo T, Ruiz A, Acuna I, Nieto-Ruiz A, Dieguez E, Sepulveda-Valbuena N, Escudero-Marin M, Garcia-Santos JA, Garcia-Ricobaraza M, Herrmann F, Moreno-Munoz JA, De Castellar R, Jimenez J, Suarez A, Campoy C. A synbiotics, long chain polyunsaturated fatty acids, and milk fat globule membranes supplemented formula modulates microbiota maturation and neurodevelopment. Clin Nutr. 2022 Aug;41(8):1697-1711. doi: 10.1016/j.clnu.2022.05.013. Epub 2022 May 23. PMID 35777109
- [Derived] Nieto-Ruiz A, Garcia-Santos JA, Verdejo-Roman J, Dieguez E, Sepulveda-Valbuena N, Herrmann F, Cerdo T, De-Castellar R, Jimenez J, Bermudez MG, Perez-Garcia M, Miranda MT, Lopez-Sabater MC, Catena A, Campoy C. Infant Formula Supplemented With Milk Fat Globule Membrane, Long-Chain Polyunsaturated Fatty Acids, and Synbiotics Is Associated With Neurocognitive Function and Brain Structure of Healthy Children Aged 6 Years: The COGNIS Study. Front Nutr. 2022 Mar 9;9:820224. doi: 10.3389/fnut.2022.820224. eCollection 2022. PMID 35356726
- [Derived] Sepulveda-Valbuena N, Nieto-Ruiz A, Dieguez E, Herrmann F, Escudero-Marin M, De-Castellar R, Rodriguez-Palmero M, Miranda MT, Garcia-Santos JA, Bermudez MG, Campoy C. Growth patterns and breast milk/infant formula energetic efficiency in healthy infants up to 18 months of life: the COGNIS study. Br J Nutr. 2021 Dec 28;126(12):1809-1822. doi: 10.1017/S000711452100057X. Epub 2021 Feb 19. PMID 33602357